CLINICAL TRIAL: NCT04724460
Title: Optimal Duration of Anticoagulation Therapy for Low-risk Pulmonary Embolism Patients With Cancer
Acronym: ONCO PE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Collaborators: Bayer Yakuhin, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Study Statistician, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0081
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Venous Thrombosis; Neoplasms; Anticoagulants
Keywords: Venous Thrombosis; Neoplasms; Anticoagulants
MeSH Terms: conditions — Venous Thrombosis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long DOAC (Active Comparator): Administration of Rivaroxaban for 18 months
  Interventions: Drug: Long DOAC
- Short DOAC (Active Comparator): Administration of Rivaroxaban for 6 months
  Interventions: Drug: Short DOAC

INTERVENTIONS:
Drug: Long DOAC — Administration of Rivaroxaban for 18 months
  Arms: Long DOAC
Drug: Short DOAC — Administration of Rivaroxaban for 6 months
  Arms: Short DOAC

SUMMARY:
The primary purpose of this study is to determine the optimal duration of anticoagulation therapy (6 months versus 18 months) with direct oral anticoagulant (DOAC) for cancer-associated low-risk pulmonary embolism patients. The major secondary purpose of this study is to investigate whether home treatment of cancer-associated low-risk pulmonary embolism patients with rivaroxaban is feasible, effective, and safe through an observational management study.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE), including pulmonary embolism (PE) and deep vein thrombosis (DVT), is a major health problem in the world. There have been many clinical studies evaluating VTE, although data on low-risk PE, including incidental PE and asymptomatic PE has been quite limited. However, low-risk PE was reported to account for a large proportion of all the diagnoses of PE detected on computed tomography in daily clinical practice, and optimal management strategies for these patients are becoming clinically more relevant. The current American College of Chest Physicians (ACCP) guidelines weakly suggest the same approach for low-risk PE patients with cancer as other PE patients with cancer. However, whether anticoagulation therapy should be continued indefinitely remains uncertain and the duration of treatment in these patients might vary widely in daily clinical practice. Recently, some observational studies reported that low-risk patients with cancer have a high risk of VTE recurrence, suggesting the benefit of prolonged anticoagulation therapy. In this open-label, superiority trial, the investigators randomly assign low-risk PE patients with active cancer to receive either rivaroxaban for 6 months (short DOAC group) or rivaroxaban for 18 months (long DOAC group).

ELIGIBILITY:
Inclusion Criteria:

* Patients with active cancer (solid and hematologic malignancies) presenting with objectively newly confirmed pulmonary embolism who are scheduled to be treated by anticoagulation therapy.
* Patients with an simplified Pulmonary Embolism Severity Index (PESI) score of 1 or less

Exclusion Criteria:

* Contraindicated patients for rivaroxaban (Clinically significant liver disease, Bacterial endocarditis, Active bleeding, Inadequate contraceptive measures if of childbearing potential, Concomitant use of strong cytochrome P-450 3A4 inhibitors or inducers or P-glycoprotein inhibitors or inducers)
* Expected life expectancy <6 months
* Patients who do not provide written informed consent
* Patients who judged to be inappropriate for enrolment by the physician (including patients at a high risk of gastrointestinal or genitourinary bleeding)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
VTE recurrence event Venous thromboembolism (VTE) recurrence event | 18 months
  VTE recurrence event is defined as pulmonary embolism (PE) and/or deep vein thrombosis (DVT) by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy.

SECONDARY OUTCOMES:
Major bleeding event (ISTH criteria) | 3 months
  Major bleeding is defined as International Society of Thrombosis and Hemostasis (ISTH) major bleeding, which consisted of a reduction in the hemoglobin level by at least 2 g/dL, transfusion of at least 2 units of blood or symptomatic bleeding in a critical area or organ.
PE-related death event | 3 months
  PE-related death event is defined as death due to a documented PE (either an objective test prior to death of the subject or PE detected during autopsy) or unexplained death (i.e. death without a clear alternate cause and not a primary consequence of subject's underlying cancer).
A composite of PE-related death, symptomatic recurrent VTE, and major bleeding (ISTH criteria) | 3 months
  PE-related death event is defined as death due to a documented PE or unexplained death. Symptomatic VTE recurrence event is defined as PE and/or DVT with symptoms accompanied by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy. Major bleeding is defined as International Society of Thrombosis and Hemostasis (ISTH) major bleeding, which consisted of a reduction in the hemoglobin level by at least 2 g/dL, transfusion of at least 2 units of blood or symptomatic bleeding in a critical area or organ.
Symptomatic VTE recurrence event | 3 months
  Symptomatic VTE recurrence event is defined as PE and/or DVT with symptoms accompanied by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy.
Hospitalization for VTE recurrence or clinically relevant bleeding events | 3 months
  Hospitalization for VTE recurrence or bleeding events. VTE recurrence event is defined as PE and/or DVT by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy. Bleeding events are clinically relevant bleeding events, which is defined as major or clinically relevant non-major bleeding. Major bleeding is defined as International Society of Thrombosis and Hemostasis (ISTH) major bleeding, which consisted of a reduction in the hemoglobin level by at least 2 g/dL, transfusion of at least 2 units of blood or symptomatic bleeding in a critical area or organ. Clinically relevant non-major bleeding event is defined as overt bleeding (i.e. is symptomatic or visualized by examination) which is not meeting the criteria for major bleeding, requires medical attention or is associated with discomfort for the subject such as pain, or impairment of activities of daily life.
Major bleeding event (ISTH criteria) | 18 months
  Major bleeding is defined as International Society of Thrombosis and Hemostasis (ISTH) major bleeding, which consisted of a reduction in the hemoglobin level by at least 2 g/dL, transfusion of at least 2 units of blood or symptomatic bleeding in a critical area or organ.
PE-related death event | 18 months
  PE-related death event is defined as death due to a documented PE (either an objective test prior to death of the subject or PE detected during autopsy) or unexplained death (i.e. death without a clear alternate cause and not a primary consequence of subject's underlying cancer).
Symptomatic VTE recurrence event | 18 months
  Symptomatic VTE recurrence event is defined as PE and/or DVT with symptoms accompanied by confirmation of new thrombus or exacerbation of the thrombus by objective imaging examinations or autopsy.
Clinically relevant non-major (CRNM) bleeding | 18 months
  A bleeding event will be classified as a clinically relevant non-major bleeding event if it is overt (i.e. is symptomatic or visualized by examination) not meeting the criteria for major bleeding, requires medical attention or is associated with discomfort for the subject such as pain, or impairment of activities of daily life.
Clinically relevant bleeding | 18 months
  Clinically relevant bleeding is defined as major or CRNM bleeding.
All-cause death | 18 months
  Death from any cause.
Bleeding-related death event | 18 months
  Bleeding-related death event is defined as a bleeding event directly led to death. Examples of fatal bleeding events are an intracranial hemorrhage that led to herniation of the brain and death within 24 hours, and a massive gastrointestinal hemorrhage that results in shock, hemodynamic collapse, and death.
Any adverse outcomes during invasive procedures | 18 months
  Adverse outcomes include bleeding events, recurrent VTE events, all-cause deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamashita Y, Morimoto T, Muraoka N, Shioyama W, Chatani R, Shibata T, Nishimoto Y, Ogihara Y, Doi K, Oi M, Shiga T, Sueta D, Kim K, Tanabe Y, Koitabashi N, Takada T, Ikeda S, Nakagawa H, Tsukahara K, Shoji M, Sakamoto J, Hisatake S, Ogino Y, Fujita M, Nakanishi N, Dohke T, Hiramori S, Nawada R, Kaneda K, Ono K, Kimura T; ONCO PE Trial Investigators. Rivaroxaban for 18 Months Versus 6 Months in Patients With Cancer and Acute Low-Risk Pulmonary Embolism: An Open-Label, Multicenter, Randomized Clinical Trial (ONCO PE Trial). Circulation. 2025 Mar 4;151(9):589-600. doi: 10.1161/CIRCULATIONAHA.124.072758. Epub 2024 Nov 18. PMID 39556015